CLINICAL TRIAL: NCT06963996
Title: Psychosocial Determinants of Sleep Health Among University Students: Implementation of a Psychoeducational Intervention
Brief Title: Efficacy of a Psychoeducational Intervention to Improve Sleep Health Among University Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, Charles M. Morin, Professor, Laval University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2023-092
Record Dates: First submitted 2025-03-18; First posted 2025-05-09 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Psychoeducational; Psychoeducational Waitlist Control
Keywords: psychoeducation; sleep; sleep hygiene; randomized controlled trial; waiting lists; control groups; sleep health; health education; intention; behavioral intention; health behavior; self-management
MeSH Terms: conditions — Sleep Hygiene; Health Education; Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): Participants assigned to the intervention group will receive first the intervention. They will complete various assessment at baseline (T0), post-intervention after the 3 weeks of intervention (T1), and 3 months after the end of the intervention (T2).
  Interventions: Behavioral: Sleep health education
- Waitlist control group (Experimental): Participants assigned to the waitlist control group complete a baseline assessment (T0), a second assessment after 3 weeks of waiting (T1), and then receive the intervention. They are assessed again after the intervention (T2) and at 3-month follow-up (T3). This design allows for pre- and post-intervention comparisons while ensuring delayed access to the program.
  Interventions: Behavioral: Sleep health education

INTERVENTIONS:
Behavioral: Sleep health education — The intervention consists of three structured sessions delivered over three weeks, with additional online follow-ups. Each session lasts 1.5 hours and takes place in the evening, with a one-week interval between sessions.
  Session 1 focuses on providing fundamental knowledge about sleep health. Session 2 introduces behavioral strategies to improve sleep health and asks participants to implement behavior change intentions.
  Session 3 reviews the implementation of the intention, the changes made or not, and addresses the relationship between stress and sleep, along with coping strategies.

SUMMARY:
This study aims to evaluate the efficacy of a psychoeducational intervention targeting the determinants of university students' sleep health. It is conducted as part of a doctoral research project.

The intervention consists of three structured sessions delivered over three weeks, with additional online follow-ups. Each session lasts 1.5 hours and takes place in the evening, with a one-week interval between sessions.

Session 1 focuses on providing fundamental knowledge about sleep health. Session 2 introduces behavioral strategies to improve sleep health and asks participants to implement behavior change intentions.

Session 3 reviews the implementation of the intention, the changes made or not, and addresses the relationship between stress and sleep, along with coping strategies.

Participants are required to complete online questionnaires and a sleep diary at multiple time points: before the intervention, immediately after, and up to three months post-intervention. These assessments measure sleep habits, beliefs about sleep, and mental health indicators.

Participants are randomly assigned to one of two groups:

Intervention group, which receives the psychoeducational program first. Waitlist control group, which completes an additional follow-up before receiving the intervention.

The study design allows for a controlled evaluation of the intervention's impact on sleep-related behaviors and mental health outcomes.

DETAILED DESCRIPTION:
A process evaluation will be conducted immediately after the 3 weeks intervention to assess participants' comprehension, adherence to the intervention, as well as the accessibility and relevance of intervention content. Moreover, in terms of logistics, this involves evaluating the premises used, the facilitator, the size of the group, the number and length of sessions, the face-to-face offer, and the use of teaching aids such as manuals during the sessions. These data are collected to inform potential improvements in future iterations of the intervention and are not included as outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Students registered at Université Laval (either part-time or full-time)
* Aged between 18-30 years old
* With or without any sleep difficulties

Exclusion Criteria:

* Use of prescription sleep medication
* Diagnosed medical condition (diabetes, cancer, cardiovascular disease, chronic pain, etc.)
* Currently with a suicidal risk

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 92 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-08-03 (Actual); Study Completion 2025-08-03 (Actual)

PRIMARY OUTCOMES:
RU-SATED | Intervention group: T0 (day 1), T1 week 4 (post 3 weeks intervention), T2 week 16 (3 months post-intervention). Waitlist control group: T0 (day 1), T1 (3 weeks later T0), T2 week 8 (post 3 weeks intervention), T3 week 20 (3 months post-intervention).
  RU-SATED is the instrument used to measure sleep health. Sleep health varies according to individual, social and environmental conditions, and emphasises that good sleep is not simply the result of an absence of sleep disorders. In terms of its components, sleep health relates to (1) sleep duration, or the total number of hours of sleep obtained over 24 hours, (2) sleep efficiency, corresponding to the ease or otherwise with which an individual falls asleep and returns to sleep, and (3) timing, or how our sleep fits into a 24-hour day, (4) alertness, or sleepiness, which concerns a person's ability to maintain a state of attentive wakefulness throughout the day, (5) satisfaction, or subjectively represented sleep quality, and finally (6) sleep regularity.
  More specifically, RU-SATED score is distributed between 0 and 12, with the higher the score, the better the person's sleep health.
Sleep satisfaction | 1-week daily self-reports at each time point: T0 (day 1), T1 week 4 (post 3-week intervention), T2 week 16 (3-month follow-up); waitlist group: T0, T1 (3 weeks later), T2 week 8 (post 3-week intervention), T3 week 20 (3-month follow-up).
  Sleep satisfaction will be assessed using a single-item question from a sleep diary completed by participants each morning for seven consecutive days. The item reads: "How would you rate the quality of your sleep?" Responses are recorded on a 5-point Likert scale ranging from 1 ("very restless") to 5 ("Very deep"). Daily scores will be summed to obtain a total sleep satisfaction score ranging from 7 to 35. Higher scores indicate a higher perceived sleep quality. The measure provides a subjective evaluation of sleep quality from the participant's perspective.
Sleep timing | 1-week daily self-reports at each time point: T0 (day 1), T1 week 4 (post 3-week intervention), T2 week 16 (3-month follow-up); waitlist group: T0, T1 (3 weeks later), T2 week 8 (post 3-week intervention), T3 week 20 (3-month follow-up).
  Self-reported bedtime and wake-up time recorded daily in a sleep diary. Used to calculate the timing of sleep onset and wake time, as well as midpoint of sleep.
Sleep efficiency | 1-week daily self-reports at each time point: T0 (day 1), T1 week 4 (post 3-week intervention), T2 week 16 (3-month follow-up); waitlist group: T0, T1 (3 weeks later), T2 week 8 (post 3-week intervention), T3 week 20 (3-month follow-up).
  Calculated from self-reported sleep diary entries as the ratio of total sleep time to time in bed, expressed as a percentage.
Sleep duration | 1-week daily self-reports at each time point: T0 (day 1), T1 week 4 (post 3-week intervention), T2 week 16 (3-month follow-up); waitlist group: T0, T1 (3 weeks later), T2 week 8 (post 3-week intervention), T3 week 20 (3-month follow-up).
  Self-reported total sleep time calculated daily using sleep onset and wake-up time entries in the sleep diary.
Sleep regularity | 1-week daily self-reports at each time point: T0 (day 1), T1 week 4 (post 3-week intervention), T2 week 16 (3-month follow-up); waitlist group: T0, T1 (3 weeks later), T2 week 8 (post 3-week intervention), T3 week 20 (3-month follow-up).
  Measured via self-reported bedtimes and wake-up times across multiple days using a sleep diary. Variability will be calculated using the standard deviation of sleep and wake times to assess sleep regularity.

SECONDARY OUTCOMES:
Sleep hygiene beliefs | Intervention group: T0 (day 1), T1 week 4 (post 3 weeks intervention), T2 week 16 (3 months post-intervention). Waitlist control group: T0 (day 1), T1 (3 weeks later T0), T2 week 8 (post 3 weeks intervention), T3 week 20 (3 months post-intervention).
  This outcome is assessed students' beliefs about sleep hygiene using the Theory of Planned Behavior (TPB). Since no standardized tools exist, items were developed based on prior research and theoretical guidelines. Validity was confirmed through factor analysis and internal consistency testing.
  The instrument includes 7-point Likert scales measuring:
  Attitudes (6 items) - Perceptions of sleep hygiene. Higher scores indicate more favorable attitudes (score range of 6 to 42).
  Subjective norms (4 items) - Perceived social expectations. Higher scores reflect stronger norms (score range of 4 to 28).
  Motivation to comply (4 items) - Importance given to others' opinions (score range of 4 to 28).
  Perceived control (4 items) - Confidence in maintaining good sleep habits (score range of 4 to 28).
  Intention (3 items) - Readiness to adopt healthy sleep behaviors (score range of 3 to 21).
  This structured approach ensures a comprehensive assessment of beliefs and behavioral influences.
Sleep Hygiene Practice Scale | Intervention group: T0 (day 1), T1 week 4 (post 3 weeks intervention), T2 week 16 (3 months post-intervention). Waitlist control group: T0 (day 1), T1 (3 weeks later T0), T2 week 8 (post 3 weeks intervention), T3 week 20 (3 months post-intervention).
  Sleep hygiene is measured by the Sleep hygiene practice scale (SHPS), which is an instrument that measures sleep hygiene including 4 domains: (1) factors related to the sleep-wake cycle (e.g. irregular bedtime/rising time, lack of exposure to outside light), (2) factors related to activation and activating behaviours (e.g. falling asleep watching television or listening to music, intense exercise in the 2 hours before going to sleep), (3) factors related to consumption and diet (e.g.going to bed hungry, drinking alcohol close to bedtime), and (4) factors related to the sleep environment (e.g. sleeping environment too noisy, too bright, too hot). The total score is distributed between 30 and 180, where the higher the score, the higher the frequency of poor sleep hygiene practices.
Self-efficacy | Intervention group: T0 (day 1), T1 week 4 (post 3 weeks intervention), T2 week 16 (3 months post-intervention). Waitlist control group: T0 (day 1), T1 (3 weeks later T0), T2 week 8 (post 3 weeks intervention), T3 week 20 (3 months post-intervention).
  This study evaluates self-efficacy in adopting, maintaining, and recovering sleep habits. Inspired by prior research, the instrument includes:
  Adoption efficacy (2 items) - Confidence in changing sleep habits despite difficulties.
  Maintenance efficacy (4 items) - Ability to sustain new sleep routines over time.
  Recovery efficacy (3 items) - Capacity to resume habits after interruption. Each item is rated on a 4-point Likert scale (1 = "Completely false," 4 = "Completely true").
  The range of scores is 2 to 8, 4 to 16 and 3 to 12 respectively. Higher scores indicate stronger self-efficacy in each domain.

OTHER OUTCOMES:
Perceived stress | Intervention group: T0 (day 1), T1 week 4 (post 3 weeks intervention), T2 week 16 (3 months post-intervention). Waitlist control group: T0 (day 1), T1 (3 weeks later T0), T2 week 8 (post 3 weeks intervention), T3 week 20 (3 months post-intervention).
  Perceived stress is evaluated using the Perceived Stress Scale (PSS), which measures how stressful life situations are perceived. This self-administered questionnaire consists of 14 items, rated on a 5-point Likert scale (0 = "Never", 1 = "Almost never", 2 = "Sometimes", 3 = "Fairly often", 4 = "Very often"). The total score ranges from 0 to 56, with higher scores indicating greater perceived stress. The PSS will be used to control for stress levels during evaluation phases, especially around exam periods, when participants are expected to report higher stress levels.
Anxiety | Intervention group: T0 (day 1), T1 week 4 (post 3 weeks intervention), T2 week 16 (3 months post-intervention). Waitlist control group: T0 (day 1), T1 (3 weeks later T0), T2 week 8 (post 3 weeks intervention), T3 week 20 (3 months post-intervention).
  Anxiety is evaluated using the GAD-7 (Generalized Anxiety Disorder scale). This 7-item self-report tool assesses anxiety symptoms experienced over the past two weeks, such as feeling nervous, unable to control worries, or having difficulty relaxing. Each item is scored from 0 to 3, indicating the frequency of symptoms. The total score ranges from 0 to 21, with thresholds at 5, 10, and 15 categorizing anxiety as mild, moderate, or severe. A score of 10 or higher is used to identify clinical levels of anxiety, which will be applied to distinguish students with clinically significant anxiety in this study.
Depression | Intervention group: T0 (day 1), T1 week 4 (post 3 weeks intervention), T2 week 16 (3 months post-intervention). Waitlist control group: T0 (day 1), T1 (3 weeks later T0), T2 week 8 (post 3 weeks intervention), T3 week 20 (3 months post-intervention).
  The PHQ-9 will assess students' depression levels, with scores ≥10 indicating clinical depression. This self-administered questionnaire evaluates the presence and severity of depressive symptoms over the past two weeks. It consists of nine items rated on a four-point Likert scale (0 = "not at all" to 3 = "nearly every day"), resulting in a total score from 0 to 27. Severity thresholds are: minimal (1-4), mild (5-9), moderate (10-14), moderately severe (15-19), and severe (20-27).
Insomnia Severity Index | Intervention group: T0 (day 1), T1 week 4 (post 3 weeks intervention), T2 week 16 (3 months post-intervention). Waitlist control group: T0 (day 1), T1 (3 weeks later T0), T2 week 8 (post 3 weeks intervention), T3 week 20 (3 months post-intervention).
  The Insomnia Severity Index (ISI) assesses nocturnal and daytime insomnia symptoms. It consists of seven items rated on a five-point Likert scale, with total scores ranging from 0 to 28. Clinical thresholds categorize scores as no insomnia (0-7), subclinical insomnia (8-14), moderate clinical insomnia (15-21), and severe clinical insomnia (22-28). The ISI is a validated and reliable tool (Cronbach's alpha = .74). This measure will be used to control for sleep health outcomes, distinguishing students with scores above 10, indicating probable insomnia.
Sociodemographic measures | Day 1 (T0)

CONTACTS AND LOCATIONS:
Locations (1):
- Centre d'études des troubles du sommeil (CETS), Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No